CLINICAL TRIAL: NCT04243642
Title: PJ-011726 IntelliSpace Cognition MCI Study
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Qserve (Industry); Dent Neurologic Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ICBE-2-34585
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: MCI; Cognitive Function 1, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: IntelliSpace Cognition — Philips IntelliSpace Cognition (ISC) is a digital assessment platform that supports Healthcare Professionals (HCP) in assessing the cognition of individuals. It consists of two interfaces connected to the DCDx-module in the cloud. ISC is hosted on the Philips Health Suite Digital Platform (HSDP). The first interface is the patient's interface and is presented via a tablet to collect data on how the patient performs a series of tests. The second interface is the clinician's interface and can be used on any PC or tablet. It allows for assessments to be selected and administered, observations made, data analytics performed and the generation of a report.

SUMMARY:
This study aims to create a reference database of digital cognitive assessment data in combination with neuroimaging data of patients with mild cognitive impairment. The investigators will explore and derive correlations between parameters from routine MRI images and brain volumetric analysis and the digital cognitive data to identify parameters that are relevant to classify MCI patients vs preexisting healthy control data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-80
2. Patient is able to give consent
3. MCI or amnestic MCI diagnosis by a clinical specialist, such as a neurologist - diagnosis not older than 12 months prior to inclusions date.
4. If 3D T1 MRI images are present they cannot be older than 6 months prior to the MCI clinical diagnosis was made.
5. Must be proficient in American English.
6. If patient has vision impairment or hearing loss, must be corrected to normal.
7. Must have use of fingers, hands, and arms to be able to use a pencil to write symbols.
8. Must be able to understand test instructions and participate fully in testing.

Exclusion Criteria:

1. Currently admitted to a hospital, assisted living, nursing home or a psychiatric facility.
2. Diagnosed with a (neurological) disorder other than MCI or aMCI, i.e.:

   * Current primary neurodegenerative diseases (e.g., Parkinson's disease, brain tumor, dementia)
   * Stroke
   * Current TBI
   * Current epilepsy [if # seizures ≤ 2 and not receiving ongoing treatment for seizures, and not currently seeking medical evaluation or attention related to seizures, patient can be accepted],
   * Current encephalitis
   * Current language disorder (expressive or mixed receptive/expressive excluded; articulation disorder is ok)
   * Current learning disorder
   * Current or past psychotic disorder
   * Current severe mood disorder (in the case of Major Depressive Disorder in remission or with no current episode, and Dysthymic and Adjustment disorder, examinee can be accepted)
   * Current severe anxiety disorder (e.g., PTSD, GAD, OCD) with symptoms significant enough to interfere with optimal test performance (in the case of phobias, examinee can be accepted)
   * Current or past Autism Spectrum Disorder or Intellectual Disability
   * Primarily nonverbal or uncommunicative
   * Current aphasia
   * LUPUS
   * Multiple Sclerosis
   * Sleep apnea (moderate or severe, Apnea-Hypopnea Index <15 is acceptable)
3. Major structural intracranial abnormalities and brain disorders on prior imaging study (in the last 12 months), i.e.:

   * Major developmental disorders (e.g., polymicrogyria, schizencephaly)
   * Intracranial tumors: intraaxial (brain tumors); extraaxial (tumors of bone and meninges) insofar they exert mass effect on the brain with edema or gliosis
   * Chronic brain injury and acquired focal or diffuse loss of normal parenchyma regardless of the etiology (e.g. prior stroke,brain surgery, trauma, atrophy due to neurodegenerative disease such as frontotemporal degeneration; or other causes), with the exception of age related changes (e.g. mild-moderate cerebral volume loss) on either side and prior surgery that involved only the skull but not the brain
   * Vascular encephalopathy, defined as Fazekas grade 2 or lower
4. Any history of having been unconscious related to TBI or "medical condition" > 20 minutes or have had any head-injury resulting in an overnight hospital stay
5. Any history of a medical event requiring resuscitation in which examinee was non-responsive for > 15 minutes
6. Currently receiving chemotherapy treatment, or have received chemotherapy treatment in the past 2 months
7. Any history of ECT or radiation to the CNS
8. Currently diagnosed with substance abuse or dependence, or have carried any substance abuse or dependence diagnosis in the past year (> 1 year in remission diagnoses are ok)
9. A current average alcohol consumption of 4 or more units per day. Long term alcohol abusers are excluded as well (e.g., abused substance for more than 10 years)
10. Currently taking medication that might impact test performance (i.e. anti- convulsants, antipsychotics, benzodiazepines, psychostimulants, opioids, tricyclic Antidepressants, Oxybutynin)
11. Disruptive behavior or insufficient compliance with testing to ensure a valid assessment
12. Non-valid health insurance in USA

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include N=125 patients with Mild Cognitive Impairment (MCI).
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Compare performance of patients with Mild Cognitive Impairment | Feb-2020 until Dec-2021
  Create a database of digital cognitive assessment data in combination with neuroimaging data of patients with mild cognitive impairment to: Compare performance of patients with Mild Cognitive Impairment (MCI) to normative data of the healthy US population and characterize a MCI cognitive profile.
Derive correlations between parameters | Feb-2020 until Dec-2021
  Create a database of digital cognitive assessment data in combination with neuroimaging data of patients with mild cognitive impairment to: Derive correlations between parameters derived from MRI images (NeuroQuant scores) and the digital cognitive data.
Identify (combinations of) parameters | Feb-2020 until Dec-2021
  Create a database of digital cognitive assessment data in combination with neuroimaging data of patients with mild cognitive impairment to: Identify (combinations of) parameters that are relevant to classify MCI patients vs healthy controls.
Explore predictive values | Feb-2020 until Dec-2021
  Create a database of digital cognitive assessment data in combination with neuroimaging data of patients with mild cognitive impairment to: Explore predictive value of combination of neuroimaging and digital cognitive outcome parameters to predict MCI to Alzheimer's disease conversion.

SECONDARY OUTCOMES:
Exploratory analysis to find new outcome measures from the raw input data of the digital cognitive tests. | Feb-2020 until Dec-2021
Evaluate the performance of ISC scoring algorithms. | Feb-2020 until Dec-2021
To explore usability aspects of ISC with MCI patients. | Feb-2020 until Dec-2021

CONTACTS AND LOCATIONS:
Locations (1):
- DENT Neurologic Institute, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided